CLINICAL TRIAL: NCT06928961
Title: Implementation of a Patient Portal and Tailored Patient-Reported Outcome Measures to Improve Health Problem Detection and Retention in HIV Care: The DRHIVe Study
Brief Title: A Patient Portal and PROMs to Improve Health Problem Detection and Retention in HIV Care: The DRHIVe Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Programme National de Mentorat sur le VIH et les Hépatites (PNMVH) (Unknown); Portail VIH/sida du Québec (Unknown); Assistance Publique - Hôpitaux de Paris (Other); Unité de Soutien SSA Québec (Unknown)
Responsible Party: Principal Investigator, Dr. Bertrand Lebouche, Clinician-Scientist and Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 186089_1
Record Dates: First submitted 2025-02-24; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: HIV; Patient-Reported Outcomes (PRO); Screening; Patient Portals
Keywords: HIV; Implementation; mHealth; Patient-reported outcome measures; PROMs; Screening; Patient portal; Mixed methods; Stakeholder engagement; Quebec; Canada; HIV care
MeSH Terms: interventions — Patient Portals

STUDY DESIGN:
Intervention Model Description: This is a single-site, unblinded, 24-month pragmatic trial using a hybrid type 2 implementation-effectiveness design. The intervention will be progressively rolled out at 6-month intervals, until all participants (9 physicians and 360 patients) receive it. For rollout, 9 clusters formed of 1 physician and 40 of their patients will be randomly assigned to a rollout schedule. From 0-6 months, all participants with be in the control condition. At months 6, 12, and 18, 3 distinct clusters will begin the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): In this arm, the control period will be 6 months followed by 18 months of intervention.
  Interventions: Other: Patient portal with patient-reported outcome measure administration, appointment calendar and reminders, access to lab test results, and educational material
- Arm 2 (Experimental): In this arm, the control period will be 12 months followed by 12 months of intervention.
  Interventions: Other: Patient portal with patient-reported outcome measure administration, appointment calendar and reminders, access to lab test results, and educational material
- Arm 3 (Experimental): In this arm, the control period will be 18 months, followed by 6 months of intervention.
  Interventions: Other: Patient portal with patient-reported outcome measure administration, appointment calendar and reminders, access to lab test results, and educational material

INTERVENTIONS:
Other: Patient portal with patient-reported outcome measure administration, appointment calendar and reminders, access to lab test results, and educational material — Patients in the intervention will be trained to register on and use the patient portal. The following portal features will be used and studied in this project: the appointment calendar, PROMs administration, reminders (e.g., for appointments), educational materials, and access to personal lab results. Educational materials in the portal will include information on what to expect during HIV clinic visits, how to interpret HIV lab reports, and instructional videos on using the portal. Prior to visiting their HIV physician, patients will have continuous access to several portal features (calendar, education, and lab results, if applicable), and receive reminders (within 48 hours) of their clinic appointment and to complete the PROMs. Physicians will acquire their patients' PROM scores via the patient portal and receive training on how to do so. Patients and physicians are expected to review the PROM results and consider them during each clinic visit.

SUMMARY:
Too often, people living with HIV (PLHIV) face challenges, including additional health and psychosocial problems, that complicate self-care, like medication-taking and medical appointment attendance. Healthcare providers are not always aware when patients face these difficulties. A 'patient portal' is an online application that can give patients access to their medical records, appointment reminders, and questionnaires to inform providers about their health and wellbeing. Patient portals in HIV care can help providers detect patient problems and improve care. At the McGill University Health Centre's (MUHC) HIV care service, a survey showed great interest in a patient portal among both PLHIV and healthcare providers. Yet, little is known on how best to integrate a portal in HIV care settings and ensure it is accessible to patients. This project will be conducted at the MUHC's HIV care service in Montreal, Quebec which has over 2,000 patients. Participating patients will log on to a patient portal through a smartphone application and have a calendar of their HIV care appointments, health questionnaires to complete (previously chosen by people with HIV and healthcare providers), reminders for both and access to educational material. HIV physicians will be able to see their patients' questionnaire results to discuss them during clinic appointments. The project's objectives are to better understand what is needed to successfully integrate a portal in similar HIV practices with diverse patients and learn how acceptable and usable it is for HIV patients and doctors. The project will also examine how patient portal use impacts satisfaction, attendance, and physician detection of specific health problems. Furthemore, it will consider how patient sex, age, and ethnicity influence the results. People with HIV, providers, and staff at the study site will be involved in decision-making about this project. Over its 5-year duration, knowledge will be gained and shared on how to expand portal use efficiently and equitably in similar HIV care centers.

DETAILED DESCRIPTION:
Background HIV care involves challenges; people living with HIV (PLHIV) face greater risks of several comorbidities and psychosocial difficulties, which often impede medication adherence, appointment attendance, and other aspects of HIV self-management. For providers, detection of many of these issues (e.g., symptoms, depression, substance use) largely relies on patients reporting them and they may go untreated. Evidence shows that patient portals and patient-reported outcome measures (PROMs) can help improve HIV management. How best to implement and ensure equitable access to these tools is less clear.

Aims This project will deploy a patient portal with a standard set of PROMs previously chosen through HIV stakeholder consultations led by the research team (PLHIV, healthcare professionals…). The study site, the Chronic Viral Illness Service (CVIS) of the McGill University Health Centre, serves over 2,000 PLHIV and is the largest university hospital-based HIV center in Montreal, Quebec. The study trial will assess an implementation strategy and patient and physician perceptions of the intervention (Aim 1) and evaluate the effectiveness of available portal functions (patient lab results, appointment calendar, PROMs, reminders, educational material) in improving health service and patient outcomes (Aim 2). HIV stakeholders will be engaged throughout this 5-year project, with representation of underserved HIV communities.

Methods A single-site, multi-method, 24-month unblinded trial will be led, with a hybrid type 2 effectiveness-implementation design and progressive intervention roll-out to all participants. Nine HIV physicians will participate with 360 of their patients, setting targets for sex, age, and race/ethnicity (factors tied to differential portal use). Patients will be trained to use the portal. Appointment and PROMs-completion reminders will be automated. Patients receiving the intervention will fill out PROMs prior to meeting their HIV physician at 6-month intervals. Physicians will be trained to consult the data via an online dashboard.

For Aim 1, study questionnaires (every 6 months), will assess patient and physician satisfaction with the intervention and perceived acceptability and usability. Portal metadata, trial data (e.g., recruitment rate) and qualitative data (e.g., semi-structured interviews, coordinator fieldnotes, meeting minutes) will be analyzed, in part, to determine fidelity and feasibility. For Aim 2, outcomes will be measured every six months. Patient outcomes include satisfaction with care and medical appointment attendance which will be based on questionnaire data and study site data, respectively. Service outcomes include physician detection of health-related problems screened for with the PROMs and patient-centered care which will be obtained from physician consultation notes and questionnaire data, respectively. Data will be analyzed, in part, with an implementation framework (NASSS) and attend to equity. The engagement approach used includes an executive committee with patient-partners and physician-champions, and a patient advisory committee. The multidisciplinary research team includes experts in all relevant areas, including implementation science.

Expected outcomes This project will build knowledge on how to implement portals and PROMs efficiently and inclusively in similar HIV centers while potentially benefiting thousands of PLHIV at the CVIS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed living with HIV
* Adult (at least 18 years old)
* Literate in English or French
* Patient at the study site

Exclusion Criteria:

* Cognitive impairment or medical instability that prevents participation
* Insufficient mastery of French or English to participate (e.g., complete PROMs, study questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention | During the intervention at months 6, 12, 18, and 24
  Acceptability of the intervention is the primary implementation outcome. It will be measured with the Acceptability E-Scale. The minimum and maximum scores on this measure are 6 and 30, respectively, where higher scores mean greater acceptability.
Satisfaction with care | At baseline, then at months 6, 12, 18 and 24
  Satisfaction with care will be the primary effectiveness outcome measure. It will be assessed with the Short Assessment of Patient Satisfaction (SAPS) measure. The minimum and maximum scores on this measure are 0 and 28, respectively, where higher scores mean greater levels of patient satisfaction.

SECONDARY OUTCOMES:
Technology usability -Ease of use | During the intervention at months 6, 12, 18, and 24
  Technology usability is a secondary outcome for assessing the implementation. It will be measured in terms of Perceived ease of use (1 item, Single Ease Question). The minimum and maximum scores on this measure are 1 and 7, respectively, where higher scores mean greater ease of use.
Technology usability -Perceived usefulness | During the intervention at months 6, 12, 18, and 24
  Technology usability is a secondary outcome for assessing the implementation. It will be measured in terms of Perceived usefulness. The minimum and maximum scores on this measure are 1 and 7, respectively, where higher scores mean greater perceived usefulness.
Technology usability -Attitude | During the intervention at months 6, 12, 18, and 24
  Technology usability is a secondary outcome for assessing the implementation. It will be measured in terms of Attitude (likelihood to recommend the intervention). The minimum and maximum scores on this measure are 1 and 5, respectively, where higher scores mean a greater likelihood to recommend. Scores will be used to calulate the percentage of participants who are likely to recommend the intervention.
Feasibility of the intervention -Consent rate | At baseline
  Feasibility will be assessed to evaluate the implementation. It will be measured in terms of the Consent rate (the percentage of participants who consented amongst those who were eligible and approached).
Feasibility of the intervention -Retention rate | From baseline to 24 months
  Feasibility will be assessed to evaluate the implementation. It will be measured in terms of the participant Retention rate (the percentage of participants who enrolled in the study and completed the trial).
Fidelity of the intervention -PROM completion by patients | During the intervention at months 6, 12, 18, and 24
  Fidelity will be assessed to evaluate the implementation. It will be measured in terms of the percentage of visits patients completed the PROMs on time.
Fidelity of the intervention -PROM data reviewed by providers | During the intervention at months 6, 12, 18, and 24
  Fidelity will be assessed to evaluate the implementation. It will be measured in terms of the percentage of visits providers reviewed their patients' PROM results on time.
Patient management -Provider detection of PROM-related problems | At baseline, then at months 6, 12, 18 and 24
  Patient management is a secondary effectiveness outcome. It will be measured based on the detection (or not) of each health or psychosocial problem targeted by the administered PROMs, as recorded in the physician clinical notes of participating patients.
Patient-centered care | At baseline, then at months 6, 12, 18 and 24
  Patient-centered care is a secondary effectiveness outcome. It will be measured with the Health care process subscale (8 items) of the Revised Patient Perception of Patient-Centeredness Questionnaire (PCCC-R).The minimum and maximum scores on this measure are 1 and 4, respectively, where higher scores mean a less patient-centered health care process.
Self-management -Appointment attendance | At baseline, then at months 6, 12, 18 and 24
  Self-management is a secondary effectiveness outcome. It will be measured in terms of the number of patients attending appointments per the study schedule, based on study site administrative data.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand P Lebouché, MD, PhD, Principal Investigator — Department of Family Medicine, McGill University
Locations (1):
- Chronic Viral Illness Service, Division of Infectious Disease, Department of Medicine, McGill University Health Centre - Glen Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
No plan is yet in place. However, we do not exclude the possibility of eventually making the protocol, ICFs, datasets, data collection tools, etc. publicly available.

REFERENCES:
- [Background] Engler K, Lessard D, Lacombe K, Palich R, Lebouche B. Development of a core patient-reported outcome set for use in HIV care at the individual patient level in Montreal: protocol for a two-phased multimethod project. BMJ Open. 2025 Jan 15;15(1):e088822. doi: 10.1136/bmjopen-2024-088822. PMID 39819929